CLINICAL TRIAL: NCT06297317
Title: Longitudinal Changes in Achilles Tendon and Medial Gastrocnemius Muscle Architecture During a 156-km Ultradistance Trail Running Event
Acronym: Trailstiff
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Trailstiff
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-02

CONDITIONS: Achilles Tendinopathy; Calf Injury; Sport Injury; Lower Limb Injury
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experienced long-distance trail runners: All the participants of the First 'Trail Scientifique de Clécy 2021". This was a multidisciplinary protocol to investigate the mechanisms that contribute to performance during an ultradistance trail race (156-km)
  Interventions: Diagnostic Test: Ultrasound measurement of triceps surae muscle-tendon architecture

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement of triceps surae muscle-tendon architecture — The resting plantar-flexors MTU architecture assessment was performed using a conventional B-mode and extended-field-of-view (EFOV) ultrasound imaging. Achille tendon cross-sectionnal area, Medial gastrocnemius thickness, pennation angle, fascicle length and muscle length were collected on the dominant lower limb.

SUMMARY:
This study aimed to assess the longitudinal changes in triceps surae muscle-tendon architecture to an ultra distance trail running. Experienced trail runners (N=55, 78% men, age: 45.2 [13.5] years) participated in a 156-km trail run (6000m climbing) consisting in six 26-km laps. The resting architectural properties of triceps surae muscle-tendon were measured using ultrasound imaging for Achille tendon cross-sectional area (AT CSA), medial gastrocnemius muscle pennation angle, thickness, length and fiber length. Measurements were performed the day before the race (Baseline), at 52-km (T1), at 104-km (T2), at 156-km (T3) and 12 hours after the race (H12).

ELIGIBILITY:
Inclusion criteria

* Experienced runners voluntarily participating in the Trail Scientifique de Clécy (156 km/6000 D+)
* Participants who had already completed 2 ultratrail races (+160 km and -160 km), at least one of them in the past 24 months; the participants had to justify their events and rankings
* Participants affiliated with a social security system or those who were a beneficiary of such a system
* Participants who could speak and read the French language
* Participants with the ability to physically participate in the ultraendurance race
* Participants with the ability to provide written consent for participation in the study

Exclusion criteria

* Participants with cardiac or extracardiac contraindications to intense physical activity
* Participants who had run a mountain ultramarathon (160 km) after September 2, 2021
* Pregnant or breastfeeding women
* Minor participants
* Participants included in another biomedical research protocol during this study
* Participants with recent muscular and orthopedic injuries, limiting running for <15 days
* Participants with a history of ankle joint surgery (eg, arthrodesis)
* Participants with a history of foot or ankle surgery
* Participants with lower-limb pathology or trauma

Ages: 25 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the participants engaged in the First Trail Scientifique de Clécy 2021(https://pubmed.ncbi.nlm.nih.gov/35704381/)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Achille tendon cross sectional area | Five time points: (1) at baseline, the day before the 156-km race, (2) during the race, at 52-km, (3) during the race, at 104-km, (4) immediately after the race, at 156-km and (5) at 12-hours after arrival.
  Mid-portion Achille tendon cross sectional area was measured (in mm²) using B mode ultrasound imaging
Medial gastrocnemius thickness | Five time points: (1) at baseline, the day before the 156-km race, (2) during the race, at 52-km, (3) during the race, at 104-km, (4) immediately after the race, at 156-km and (5) at 12-hours after arrival.
  Medial gastrocnemius thickness was measured at the inferior third of muscle llength (in mm) using B mode ultrasound imaging
Medial gastrocnemius pennation angle | Five time points: (1) at baseline, the day before the 156-km race, (2) during the race, at 52-km, (3) during the race, at 104-km, (4) immediately after the race, at 156-km and (5) at 12-hours after arrival.
  Medial gastrocnemius pennation angle was measured at the inferior third of muscle llength (in °) using B mode ultrasound imaging
Medial gastrocnemius fascicle length | Five time points: (1) at baseline, the day before the 156-km race, (2) during the race, at 52-km, (3) during the race, at 104-km, (4) immediately after the race, at 156-km and (5) at 12-hours after arrival.
  Medial gastrocnemius fascicle length was calculated under the assumption of linearity as Fascicle Lnegth = Muscle Thickness / sin (Pennation angle) measured at the inferior third of muscle length (calculated in mm) using B mode ultrasound imaging
Medial gastrocnemius muscle length | Five time points: (1) at baseline, the day before the 156-km race, (2) during the race, at 52-km, (3) during the race, at 104-km, (4) immediately after the race, at 156-km and (5) at 12-hours after arrival.
  Medial gastrocnemius muscle length was measured using an extended-field-of-view (EFOV) ultrasound imaging

SECONDARY OUTCOMES:
Finisher status | One time point, after the race
  Participants were classifioed as "Finishers" or "Did not finish" whether they completed the 156-km race, or not
Average speed | Four time point (1) during the race, at 52-km, (2) during the race, at 104-km, (3) during the race, at 156-km and (4) for the whole race.
  Average speed was calculated using the time per lap and distance for each lap

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauvieux B, Hingrand C, Drigny J, Hodzic A, Baron P, Hurdiel R, Jouffroy R, Vauthier JC, Pessiglione M, Wiehler A, Degache F, Pavailler S, Heyman E, Plard M, Noirez P, Dubois B, Esculier JF, Nguyen AP, Van Cant J, Roy Baillargeon O, Pairot de Fontenay B, Delaunay PL, Besnard S. Study of the Kinetics of the Determinants of Performance During a Mountain Ultramarathon: Multidisciplinary Protocol of the First Trail Scientifique de Clecy 2021. JMIR Res Protoc. 2022 Jun 15;11(6):e38027. doi: 10.2196/38027. PMID 35704381